CLINICAL TRIAL: NCT03949816
Title: The Influence of Doctor-patient Communication on Treatment Expectation, Placebo and Nocebo Response
Acronym: SENSE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Philipps University Marburg (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 2019-20k
Record Dates: First submitted 2019-05-06; First posted 2019-05-14 (Actual); Last update posted 2019-05-14 (Actual); Status verified 2019-05

CONDITIONS: Healthy Participants
Keywords: patient-centered communication; doctor-centered communication; placebo; nocebo; outcome expectation; blood pressure; heart rate; patient-physician communication

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- patient-centered communication style (Experimental): The patient-centered style is characterized by features such as empathetic communication, open questions, and uses an easily understandable language.
  Interventions: Other: medical consultation: different doctor-patient-centered style of communication
- doctor-centered communication style (Experimental): The doctor-centered style is defined by an authoritarian and goal-oriented communication. The doctor uses medical terms instead of lay language.
  Interventions: Other: medical consultation: different doctor-patient-centered style of communication
- information letter (Active Comparator): In the active control treatment participants receive all information about the herbal medical product in an information letter but have no contacted with the simulated doctor.
  Interventions: Other: information letter / no medical consultation

INTERVENTIONS:
Other: medical consultation: different doctor-patient-centered style of communication — Different doctor-patient communication
  Arms: doctor-centered communication style; patient-centered communication style
Other: information letter / no medical consultation — In the control treatment participants receive all information about the herbal medical product in an information letter but have no contacted with the simulated doctor.
  Arms: information letter

SUMMARY:
The purpose of this study is to determine whether a patient-centered compared to doctor-centered communication style of a physician influences the treatment expectation and the placebo and nocebo response in healthy individuals.

DETAILED DESCRIPTION:
Doctor-patient communication is crucial for the success of treatment and patients´ quality of life. It could be shown that the medical communication style during the consultation has an effect on the treatment expectation and can therefore positively influence the effect of a sham treatment (placebo ointment). The doctor's communication style has already been successfully manipulated in experimental designs. However, the question remains to what extent the doctor's communication style is related to the placebo/nocebo response and the change in effect-related expectations after a one-week intake of a supposedly medical herbal product (drug-free placebo).

It is expected that the patient-centered communication style of the physician has a positive impact on the reduction of stress (placebo response) and the effect-related cognitive expectations. Furthermore, the physician-centered communication style is expected to negatively impact potential side effects (nocebo response) and impact-related expectations.

Participants will be recruited via posters on public notice boards and e-mail distribution lists. After individuals register for participating in the study, they are called by a study assistant. Eligibility criteria are checked and participants are asked questions about control variables (sociodemographic data (age, sex, profession) and symptom report (Generic Assessment of Side Effects GASE)). The subjects are told that an herbal medical product (drug-free placebo pill) is tested for the reduction of stress symptoms (cover story). Subjects are randomly assigned to 3 groups (2 experimental groups: patient-centered communication style, doctor-centered communication style, control treatment: information letter). Eligible participants come in the lab for an experimental appointment. They first complete a questionnaire at baseline assessment about control variables (further sociodemographic data, disability of stress symptoms, anxiety (trait), negative and positive affectivity, communication preferences, beliefs about medicines, adherence) and outcome variables (treatment expectation, placebo response, Nocebo response, blood pressure and heart rate).

Participants in the experimental groups are then informed by a simulated doctor (played by a study assistant) about indications and side effects of the herbal medical product. The doctor applies either a patient-centered or doctor-centered communication style. The patient-centered style is characterized by features such as empathetic communication, open questions, and uses an easily understandable language. The doctor-centered style is defined by an authoritarian and goal-oriented communication. The doctor uses medical terms instead of lay language. In the control treatment participants receive all information about the herbal medical product in an information letter but have no contacted with the simulated doctor. Participating subjects, who receive a medical consultation, complete a brief questionnaire after doctor's consultation about the satisfaction with the consultation and the anticipated treatment expectancy (post-consultation). Then participants in all three groups are asked to take the herbal medical product (placebo pill). At the end of the experimental appointment, participants are asked to complete another questionnaire about the outcome variables (treatment expectation, placebo response, Nocebo response, blood pressure and heart rate) (post-intake). Participating subjects are instructed to take the placebo pill once a day over the next week. Seven days after the first appointment participants are invited to come to the lab for a follow-up assessment (1-week follow-up).

The treatment expectancy is operationalized with visual analogue scale about participant's treatment outcome expectations (VAS, see primary outcomes) at post-intake and 1-week follow-up. The placebo effect is operationalized with visual analogue scale about the relaxation level (VAS, see secondary outcomes) at post-intake and 1-week follow-up.

The nocebo effect is operationalized with the number of symptoms and symptom severity (Generic Assessment of Side Effects GASE, see secondary outcomes) attributed by participants to a medication side effect at post-intake and 1-week follow-up.

ELIGIBILITY:
Inclusion Criteria:

* female
* between 18 and 35 years
* healthy
* adequate ability to see
* fluent in German (reading and writing)

Exclusion Criteria:

* regular intake of medication that enhances relaxation
* intake of psychotropic drugs
* during the past 2 years in psychotherapeutic treatment for diagnosed mental disorder
* current pregnancy or lactation
* students enrolled in medicine, psychology or pharmacy

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-05-20 (Estimated); Primary Completion 2019-10-20 (Estimated); Study Completion 2019-11-01 (Estimated)

PRIMARY OUTCOMES:
Change in treatment outcome expectations from baseline to post-intake | Change in treatment outcome from baseline to post-intake (within 10 minutes after intake of first placebo pill)
  Visual analogue scale (VAS) measuring participant's treatment outcome expectations at baseline and at post-intake. Minimum VAS score: 0% - "the herbal medical product will not help me to reduce my stress symptoms", maximum VAS score: 100% - "the herbal medical product will help me to reduce my stress symptoms completely" (self-rating). A change score will be computed ("post-intake score" minus "baseline score"; Range of change score: -100 to +100). A higher score indicates a higher positive change in treatment outcome expectation from baseline to post-intake.

SECONDARY OUTCOMES:
Change in treatment outcome expectations from baseline to post-consultation | Change in treatment outcome from baseline to post-consultation (immediately after doctor-patient communication/information letter).
  Visual analogue scale (VAS) measuring participant's treatment outcome expectations at baseline and at post-consultation. Minimum VAS score: 0% - "the herbal medical product will not help me to reduce my stress symptoms", maximum VAS score: 100% - the herbal medical product will help me to reduce my stress symptoms completely" (self-rating). A change score will be computed ("post-consultation score" minus "baseline score"; Range of change score: -100 to +100). A higher score indicates a higher positive change in treatment outcome expectation from baseline to post-consultation.
Change in treatment outcome expectations from baseline to 1-week follow-up | Change in treatment Outcome from baseline to 1-week follow-up (after the one-week intake phase)
  Visual analogue scale (VAS) measuring participant's treatment outcome expectations at baseline and at 1-week follow-up. Minimum VAS score: 0% - "the herbal medical product will not help me to reduce my stress symptoms", maximum VAS score: 100% - the herbal medical product will help me to reduce my stress symptoms completely" (self-rating). A change score will be computed ("1-week follow-up score" minus "baseline score"; Range of change score: -100 to +100). A higher score indicates a higher positive change in treatment outcome expectation from baseline to 1-week follow-up.
Perceived ease | baseline assessment, post-intake (within 10 minutes after intake of first placebo pill), 1-week follow-up (after the one-week intake phase)
  VAS measuring perceived ease (operationalizes placebo effect). Minimum VAS score: 0% - no perceived ease, maximum VAS score: 100% - perceived absolute ease. A higher score indicates a higher perceived ease and operationalizes a higher placebo response (Score: 0% to 100%).
  VAS: "How calm inside do you feel at this moment?"
Perceived inner tension | baseline assessment, post-intake (within 10 minutes after intake of first placebo pill), 1-week follow-up (after the one-week intake phase)
  VAS measuring perceived inner tension (operationalizes placebo effect). Minimum VAS score: 0% - no perceived inner tension, maximum VAS score: 100% - perceived absolute inner tension. Inverted Item: A higher score indicates a higher perceived inner tension and operationalizes a lower placebo response (Score: 0% to 100%).
  VAS: "How tense do you feel inside at this moment?"
Perceived mental exhaustion | baseline assessment, post-intake (within 10 minutes after intake of first placebo pill), 1-week follow-up (after the one-week intake phase)
  VAS measuring perceived mental exhaustion (operationalizes placebo effect). Minimum VAS score: 0% - no perceived mental exhaustion, maximum VAS score: 100% - perceived absolute mental exhaustion. Inverted Item: A higher score indicates a higher perceived mental exhaustion and operationalizes a lower placebo response (Score: 0% to 100%).
  VAS: "How mentally exhausted do you feel at this moment?"
Score of symptom severity | post-intake (within 10 minutes after intake of first placebo pill), 1-week follow-up (after the one-week intake phase)
  Generic Assessment of Side Effects (GASE): Score of symptom severity (operationalizes nocebo effect). Minimum sum score: 0 - no symptom severity, maximum sum score: 105 - maximal symptom severity. A higher sum score indicates a higher score of symptom severity (Score: 0 to 105).
Number of symptoms which are attributed by participant for medication side effects | post-intake (within 10 minutes after intake of first placebo pill), 1-week follow-up (after the one-week intake phase)
  Generic Assessment of Side Effects (GASE): Number of symptoms which are attributed by participant for medication side effects (operationalizes nocebo effect). Minimum sum score: 0 - no symptoms, which are attributed for medication side effects, maximum sum score: 35 - maximal number of symptoms, which are attributed for medication side effects. A higher score indicates a higher Number of symptoms which are attributed by participant for medication side effects (Score: 0 to 35).
Diastolic blood pressure | baseline assessment, post-intake (within 10 minutes after intake of first placebo pill), 1-week follow-up (after the one-week intake phase)
  Diastolic blood pressure (measures by sphygmomanometer)
Systolic blood pressure | baseline assessment, post-intake (within 10 minutes after intake of first placebo pill), 1-week follow-up (after the one-week intake phase)
  Systolic blood pressure (measures by sphygmomanometer)
Heart rate | baseline assessment, post-intake (within 10 minutes after intake of first placebo pill), 1-week follow-up (after the one-week intake phase)
  Heart rate (measures by sphygmomanometer)
number of pills that have not been taken and returned | 1-week follow-up (after the one-week intake phase)
  number of pills that have not been taken and returned (operationalizes medication adherence)

CONTACTS AND LOCATIONS:
Overall Officials: Winfried Rief, PhD, Study Chair — Philipps-University Marburg, Faculty psychology, department clinical psychology
Locations (1):
- Philipps-University Marburg, Faculty psychology, department clinical psychology, Marburg, Hesse, Germany

REFERENCES:
- [Background] Bensing JM, Verheul W. The silent healer: the role of communication in placebo effects. Patient Educ Couns. 2010 Sep;80(3):293-9. doi: 10.1016/j.pec.2010.05.033. Epub 2010 Jul 17. PMID 20638817
- [Background] Czerniak E, Biegon A, Ziv A, Karnieli-Miller O, Weiser M, Alon U, Citron A. Manipulating the Placebo Response in Experimental Pain by Altering Doctor's Performance Style. Front Psychol. 2016 Jun 30;7:874. doi: 10.3389/fpsyg.2016.00874. eCollection 2016. PMID 27445878
- [Background] Epstein RM, Fiscella K, Lesser CS, Stange KC. Why the nation needs a policy push on patient-centered health care. Health Aff (Millwood). 2010 Aug;29(8):1489-95. doi: 10.1377/hlthaff.2009.0888. PMID 20679652
- [Background] Graugaard PK, Finset A. Trait anxiety and reactions to patient-centered and doctor-centered styles of communication: an experimental study. Psychosom Med. 2000 Jan-Feb;62(1):33-9. doi: 10.1097/00006842-200001000-00005. PMID 10705909
- [Background] Howe LC, Goyer JP, Crum AJ. Harnessing the placebo effect: Exploring the influence of physician characteristics on placebo response. Health Psychol. 2017 Nov;36(11):1074-1082. doi: 10.1037/hea0000499. Epub 2017 Mar 9. PMID 28277699